CLINICAL TRIAL: NCT05586646
Title: Effect of IV Alanyl Glutamine on Healing of Pressure Ulcers in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Specialized Hospital, Cairo, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1234
Record Dates: First submitted 2022-10-15; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer | interventions — alanylglutamine

STUDY DESIGN:
Intervention Model Description: This clinical trial will include 200 Egyptian Critically ill patients with bed sores equal or more than grade II selected from ward or ICU at Air Force specialized Hospital. They will be classified into 2 groups:
  * Group I: 100 critically ill patients will be enrolled on high protein diet and receiving IV alanyl Glutamine with dose 0.3 gm/kg/ day which equal 1.5 ml/kg/day of alanyl-glutamine until discharge from ICU, death (with duration of 2 weeks administration).
  * Group II: 100 critically ill patients will be enrolled on high protein diet either enteral or parenteral but not receiving any glutamine supplementations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): 100 critically ill patients will be enrolled on high protein diet either enteral or parenteral but not receiving any glutamine supplementations
- alanyl-glutamine group (Experimental): 100 critically ill patients will be enrolled on high protein diet and receiving IV alanyl Glutamine with dose 0.3 gm/kg/ day which equal 1.5 ml/kg/day of alanyl-glutamine until discharge from ICU, death (with duration of 2 weeks administration).
  Interventions: Dietary Supplement: alanyl-glutamine

INTERVENTIONS:
Dietary Supplement: alanyl-glutamine — Amino acid solution for parenteral nutrition containing dipeptide alanyl-glutamine
  Other Names: Dipeptiven
  Arms: alanyl-glutamine group

SUMMARY:
In this clinical trial, we will assess pressure ulcer healing rates in critically ill patients supplemented with IV Alanyl-Glutamine in comparison with critically ill patients not supplemented with alanyl-glutamine.

DETAILED DESCRIPTION:
This clinical trial will include 200 Egyptian Critically ill patients with bed sores equal or more than grade II selected from ward or ICU at Air Force specialized Hospital. They will be classified into 2 groups:

* Group I: 100 critically ill patients will be enrolled on high protein diet and receiving IV alanyl Glutamine with dose 0.3 gm/kg/ day which equal 1.5 ml/kg/day of alanyl-glutamine until discharge from ICU, death (with duration of 2 weeks administration).
* Group II: 100 critically ill patients will be enrolled on high protein diet either enteral or parenteral but not receiving any glutamine supplementations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pressure ulcers stage 2,3 or 4, non-healing admitted to Air force specialized hospital for more than a week.

Exclusion Criteria:

* Patients with renal impairment (GFR </= 30)
* Patients who require fluid restriction < 1 Litre/day.
* Patients with liver cirrhosis. (Child B and C)
* Length of stay< 2 weeks.
* Patients with deep tissue infection and/or requiring debridement of necrotic or sloughy tissue.
* Hemodynamically unstable patients. (On high dose of cardiac supports)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Percentage change in pressure ulcer length | 2 weeks
  Final ulcer length/original ulcer length x 100
Percentage change in pressure ulcer depth | 2 weeks
  Final ulcer depth/original ulcer depth x 100
Percentage change in pressure ulcer area | 2 weeks
  Final ulcer area/original ulcer area x 100
Percentage change in proportion of viable wound tissue | 2 weeks
  Final proportion of viable wound tissue /original proportion of viable wound tissue x 100

CONTACTS AND LOCATIONS:
Overall Officials: Enas Mogawer, Professor, Study Director — Air Force Specialized Hospital
Locations (1):
- Air Force Specialized Hospital, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No